CLINICAL TRIAL: NCT02615184
Title: A Phase 2, Double-Blind, 36-Week, Multicenter Study to Assess the Safety and Effectiveness of Daily Oral Administration of Dexlansoprazole Delayed-Release Capsules for Healing of Erosive Esophagitis (EE) and Maintenance of Healed EE in Pediatric Subjects Aged 2 to 11 Years With EE
Brief Title: A Study to Check the Safety of Dexlansoprazole and Learn If it Can Heal Erosive Esophagitis (EE) and Keep it Healed in Children 2 to 11 Years Old
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-390MR_205; 2022-501350-11-00 (EU CTIS Number: EU CTIS); U1111-1166-8811 (Registry Identifier: WHO)
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Erosive Esophagitis
Keywords: Drug therapy
MeSH Terms: interventions — Dexlansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healing Period: Dexlansoprazole 60 mg (Experimental): Dexlansoprazole 60 mg, capsules, orally, once, daily, for 8 weeks.
  Interventions: Drug: Dexlansoprazole
- Healing Period: Dexlansoprazole 30 mg (Experimental): Dexlansoprazole 30 mg, capsules, orally, once, daily, for 8 weeks.
  Interventions: Drug: Dexlansoprazole
- Maintenance of Healed EE: Dexlansoprazole 30 mg (Experimental): Participants on Dexlansoprazole 60 mg treatment arm in Healing Period will receive half dose, dexlansoprazole 30 mg, capsules, orally, once, daily, for 16 weeks in the Maintenance Period.
  Interventions: Drug: Dexlansoprazole
- Maintenance of Healed EE: Dexlansoprazole 15 mg (Experimental): Participants on Dexlansoprazole 30 mg treatment arm in Healing Period will receive half dose, dexlansoprazole 15 mg, capsules, orally, once, daily, for 16 weeks in the Maintenance Period.
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole capsules
  Other Names: Dexilant

SUMMARY:
Gastroesophageal reflux disease (GERD) is caused by food or acid coming up from the stomach into the esophagus, repeatedly. The esophagus is the tube that carries food and liquids from the mouth to the stomach. The body uses stomach acid to break down food, but when acid rises up into the esophagus it can hurt or damage it. People with GERD often feel food coming back up into the throat and mouth and have a burning feeling in their stomach, chest, or throat, called heartburn. Other symptoms of GERD include pain in the stomach or throat, difficulty eating, and throwing up. Sometimes GERD damages the lining of the esophagus, creating breaks. This is called erosive esophagitis (EE).

Dexlansoprazole is a type of medicine that helps lower the amount of acid made in the stomach. It has been shown to heal EE and maintain (keep) healing of EE in adults and teenagers. This study is being done to find out if dexlansoprazole can also heal EE and maintain the healing of EE in children.

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. Dexlansoprazole is being tested to heal EE and maintain healing of EE in pediatric participants aged 2 to 11 years. This study will look at the healing of EE followed by maintained healing of EE in children who take dexlansoprazole.

The study will be conducted in two periods; a Healing of EE Period and a Maintenance of Healed EE Period. Approximately 76 patients will be enrolled in this study. Participants will be randomly assigned (by chance, like flipping a coin) to receive dexlansoprazole 60 milligrams (mg) or dexlansoprazole 30 mg for 8 weeks during the Healing of EE Period. Following Week 8, participants will enter the Maintenance of Healed EE Period and will receive half their healing dose of dexlansoprazole, (i.e., either 30 mg, dexlansoprazole 15 mg).

All participants will be asked to take one capsule at the same time each day throughout the study. All participants will be asked to record any time they have heartburn symptoms in a diary.

Participants who complete the 16 weeks of the Maintenance of Healed EE Period (Week 24) and have maintained healing of EE as confirmed by endoscopy, will enter a Post-Treatment Follow up Period for up to 3 months after the last dose of study drug. During this period participants will continue to complete the symptom questionnaires daily in the eDiaries and return for a clinic visit each month. Participants who require an invasive procedure or treatment with a proton pump inhibitor (PPI) or histamine 2-receptor antagonist (H2RA) for gastroesophageal reflux disease (GERD)/EE will be discontinued from the Post-Treatment Follow-up Period and a Final Study Visit will be performed.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is up to 10 months. Participants will make multiple visits to the clinic including a final visit 3 months after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant (as age appropriate) and/or parent(s) or legal guardian are capable of understanding and complying with protocol requirements.
2. Prior to any study-specific procedures being performed, the appropriate screening informed consent and the assent forms (as applicable) must be signed and dated by parent(s) or legal guardian and by the participant respectively, if appropriate.
3. Has a medical history of symptoms of GERD for at least 3 months prior to Screening.
4. Has met the eDiary qualification criteria as assessed by the PGSDD, defined as hurting or burning in the stomach, chest, or throat on at least 3 of any 7 consecutive days during the Screening Period. (Note: If an endoscopy performed within 1 week of signing screening informed consent and assent [as applicable] is used to confirm diagnosis of EE, the participant does not need to meet this criterion).
5. Has endoscopic evidence of EE with Los Angeles (LA) Grade A to D based on the screening endoscopy performed either during the Screening Period or within 1 week prior to signing screening informed consent and assent (as applicable). An endoscopy that was performed within 1 week prior to signing screening informed consent and assent, as applicable, is an acceptable replacement for the Screening endoscopy if EE is documented by LA classification scale criterion previously described, protocol-required biopsies were collected and endoscopic pictures were obtained.
6. Is male or female and age 2 to 11 years, inclusive, at the time of screening informed consent.

Exclusion Criteria:

1. Has evidence of cardiovascular, pulmonary, central nervous system, hepatic, hematopoietic, renal, or metabolic disorder, severe allergy, asthma, or allergic skin rash that suggests any uncontrolled, clinically significant underlying disease or condition (other than the disease being studied), which may impact the ability of the participant to participate or potentially confound the study results.
2. Has a coexisting disease affecting the esophagus (eg, esophageal varices, scleroderma, viral or fungal infection, or esophageal stricture), history of radiation therapy or cryotherapy to the esophagus, caustic or physiochemical trauma such as sclerotherapy to the esophagus.
3. Has any findings in his/her medical history, physical examination, or safety clinical laboratory tests giving reasonable suspicion of underlying disease that might interfere with the conduct of the trial.
4. Has a history of hypersensitivity or allergies to dexlansoprazole or any component of dexlansoprazole capsules or any PPI (including lansoprazole, omeprazole, rabeprazole, pantoprazole, or esomeprazole) or antacids.
5. Is required to take excluded medications or it is anticipated that the participant will require treatment with at least 1 of the disallowed concomitant medications during the study evaluation period.
6. Has a condition that may require inpatient surgery during the course of the study.
7. Has a known history of Barrett's with dysplastic changes in the esophagus.
8. Has a known history of eosinophilic esophagitis (EoE) or histologic findings suggestive of EoE (≥15 eosinophils per high-powered field [HPF]).
9. Has history of celiac disease, tests positive for tissue transglutaminase (tTG) antibody, or has confirmed disease by histology.
10. Has history of inflammatory bowel disease, or irritable bowel syndrome.
11. Has active gastric or duodenal ulcers within 4 weeks prior to Day -1. If present >4 weeks prior to Day -1, ulcers must not be present upon screening endoscopy.
12. Requires dilatation of esophageal strictures and/or strictures preventing passage of the endoscope during the Screening endoscopy. Schatzki's ring (a ring of mucosal tissue near the lower esophageal sphincter) is acceptable.
13. A female participant who has reached menarche by Day -1.
14. Is known to be positive for the human immunodeficiency virus (HIV).
15. Has current or clinical history of Zollinger-Ellison syndrome or other hypersecretory condition.
16. Has a history of gastric, duodenal, or esophageal surgery except simple oversew of an ulcer. A history of gastric tube and/or percutaneous endoscopic gastrostomy (PEG) placement is allowed.
17. Had an acute upper gastrointestinal hemorrhage within 4 weeks prior to endoscopy.
18. Has donated or lost >10% of the total blood volume, undergone plasmapheresis, or has had a transfusion of any blood product within 90 days prior to the first dose of study drug.
19. Has a known history of alcohol abuse or illegal drug use within the past 12 months prior to the first dose of study drug.
20. Has any screening abnormal laboratory value that suggests a clinically significant underlying disease or condition that may prevent the participant from entering the study; or the participant has: creatinine >1.5 milligrams per deciliter (mg/dL), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 times the upper limit of normal (×ULN), or total bilirubin >2.0 mg/dL with AST/ALT elevated above the limits of normal values.
21. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study or may consent and assent under duress. Students of the institution/research facility who are under the supervision of, or in a subordinate role to, the investigator are also ineligible.
22. The participant, in the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.
23. Has participated in another clinical study (not including screening for Study TAK-390MR_204 [NCT02616302]) and/or has received any investigational compound within 30 days prior to Screening.
24. Tests positive for Helicobacter pylori.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Healing of EE by Week 8 | Week 8
  Healing of EE will be assessed by endoscopy.
Percentage of Participants who Maintained Healed EE from Week 8 to Week 24 | Week 8 to Week 24
  Percentage of participants who maintained healed EE from Week 8 to Week 24 among the participants who were healed at Week 8 as assessed by endoscopy.

SECONDARY OUTCOMES:
Percentage of Days Without Hurting or Burning in the Stomach, Chest or Throat Over the First 8 Weeks of Treatment | Week 8
  Daily electronic diaries (eDiaries) will be completed which contain Pediatric Gastroesophageal Reflux Disease Symptom Daily Diaries (PGSDD) questionnaires that document presence or absence of hurting or burning in the stomach, chest or throat vomiting, regurgitation and trouble eating. Parents or caregivers of participants aged 2 to 8 years will complete the PGSDD (parent) in the eDiary for their child and participants aged 9 to 11 years will complete PGSDD (child) in the eDiary themselves. The eDiaries will be completed on a daily basis reflecting a continuous 24-hour period.
Percentage of Days Without Hurting or Burning in the Stomach, Chest or Throat Over Weeks 8 to 24 Among Participants Who were Healed by Week 8 | Weeks 8 to 24
  Daily eDiaries will be completed which contain PGSDD questionnaires that document presence or absence of hurting or burning in the stomach, chest or throat vomiting, regurgitation and trouble eating. Parents or caregivers of participants aged 2 to 8 years will complete the PGSDD (parent) in the eDiary for their child and participants aged 9 to 11 years will complete PGSDD (child) in the eDiary themselves. The eDiaries will be completed on a daily basis reflecting a continuous 24-hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (25):
- United States (11):
  - University of South Alabama, Mobile, Alabama
  - University of California San Francisco, San Francisco, California
  - D&H National Research Centers, Miami, Florida
  - Children's Center for Digestive Health Care, LLC, Atlanta, Georgia
  - Gastrointestinal Associates, PA, Flowood, Mississippi
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Measurable Outcome Research, Oklahoma City, Oklahoma
  - GI for Kids, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Envision Clinical Research, LLC, Laredo, Texas
  - The Children's Hospital of The King's Daughters, Norfolk, Virginia
- Canada (2):
  - Women and Children's Health Research Institute, Edmonton, Alberta
  - London Health Sciences Centre (LHSC) - Children's Hospital, London, Ontario
- Colombia (3):
  - Hospital Universitario San Ignacio, Bogotá
  - Fundacion Valle del Lili, Cali
  - Centro Medico Imbanaco de Cali S.A, Cali
- Mexico (5):
  - Boca Clinical Trials Mexico SC, Colonia Las Americas, Mexico City
  - Inspirepharma S. de R.L. de C.V., Monterrey, Nuevo León
  - Clinical Research Institute S.C., Tlalnepantla, State of Mexico
  - El Cielo Medical Center, Puebla City
  - SMIQ S. de R.L. de C.V., Querétaro
- Poland (4):
  - In Vivo Osrodek Badan Klinicznych, Bydgoszcz, Kuyavia
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow, Lesser Poland Voivodeship
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw, Masovia
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów, Podkarpackie Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b602f4db2bf003ab49d28?idFilter=%5B%22TAK-018-2001%22%2C%22TAK-390MR_205%22%5D